CLINICAL TRIAL: NCT05235074
Title: A Clinical Study of Oncolytic Virus (OH2) Injection in the Treatment of Patients Undergoing Surgery After Recurrence of Central Nervous System Tumors
Brief Title: OH2 Oncolytic Viral Therapy in Central Nervous System Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Binhui Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BH-OH2-015
Record Dates: First submitted 2022-01-27; First posted 2022-02-10 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Central Nervous System Tumors
Keywords: Oncolytic Virus
MeSH Terms: conditions — Central Nervous System Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose escalation and dose expansion (Experimental): The dose-escalating phase of the phase I trial of OH2 injection is divided into two dose groups (10^6 CCID50/mL and 10^7 CCID50/mL).It will be administered by Ommaya reservoir injection, and the total amount of each dose in each dose group should not exceed 2ml according to the size of the tumor cavity.
  Interventions: Biological: OH2 injection

INTERVENTIONS:
Biological: OH2 injection — OH2: Oncolytic Type 2 Herpes Simplex Virus

SUMMARY:
In the first phase, it mainly explores the safety, tolerability and preliminary effectiveness of two doses of OH2 injection in the treatment of patients with recurrent central nervous system tumors; to evaluate the biodistribution and virus shedding of OH2 injection administered in the tumor cavity; to evaluate the level of anti-HSV2 antibody in patients when OH2 injection is administered intracavitary to tumor; to determine the phase II recommended dose (RP2D) of OH2 injection in the treatment of recurrent glioblastoma.

Phase IIa, to evaluate the preliminary efficacy of OH2 injection in the treatment of patients with recurrent glioblastoma after surgery, and to further evaluate the safety of OH2 in the treatment of relapsed glioblastoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, male or female;
2. Phase I trials select pathologically confirmed recurrent central nervous system tumors (including but not limited to anaplastic astrocytoma, anaplastic oligoastrocytoma, glioblastoma, gliosarcoma, anaplastic ependymoma, Medulloblastoma, malignant meningioma, melanoma, etc.) postoperative patients; Phase IIa trial selects postoperative patients with pathologically confirmed recurrent glioblastoma
3. KPS score ≥60;
4. Partial or complete tumor resection, Ommaya reservoir has been placed in the operation area, and drug administration conditions are available;
5. As assessed by the investigator, the site of injection of the trial drug is expected to be in the supratentorial area;
6. Life expectancy ≥3 months;
7. Blood routine: WBC≥ 3.0×10^9/L, ANC≥1.5×10^9/L, PLT≥100×10^9/L, Hb≥9.0 g/dL;
8. Liver and kidney function: total bilirubin ≤ 1.5 times the upper limit of the normal value; AST and ALT < 2.5 times the upper limit of the normal value; serum creatinine ≤1.5 times the upper limit of the normal value, or creatinine clearance ≥50 ml/min (calculated by Cockcroft/Gault formula);
9. Coagulation function: INR≤1.5 times the upper limit of the normal value, APTT≤1.5 times the upper limit of the normal value;
10. Women of childbearing age had a negative pregnancy test result within 14 days before enrollment. Female subjects and their spouses received effective contraceptives during and within 6 months of treatment;
11. The subjects voluntarily participated in this study, signed the informed consent form, had good compliance, and cooperated with the follow-up.

Exclusion Criteria:

1.28 days before enrollment, subjects participated in other clinical trial projects.

2.The subject has received tumor chemotherapy, targeted therapy or immunotherapy within 28 days before the first use of the test drug.

3.The subjects have received traditional Chinese medicine, modern Chinese medicine preparations and antiviral drugs within 7 days before using the test drug for the first time.

4.Subjects had received radiotherapy to the brain 3 months before their first use of the test drug.

5.Subjects with other active extracranial malignancies requiring concomitant therapy.

6.Subjects known to be allergic to the test drug or its active ingredients, excipients, and imaging contrast agents.

7.Subjects who are going to undergo or have received tissue/organ transplantation in the past.

8.The subject has active infection or unexplained fever >38.5℃ during the screening period and before the first dose.

9.Subjects with active pulmonary tuberculosis (TB) who are receiving anti-tuberculosis treatment or who have received anti-tuberculosis treatment within 1 year before screening.

10.Anti-HIV(+) or anti-HCV(+) or specific antibody (TPHA) positive or active hepatitis B (hepatitis B subjects who meet the following criteria are also eligible for inclusion: a) HBV viral load before the first dose The amount must be less than 1000 copies/ml (200 IU/ml), and subjects should receive anti-HBV treatment throughout the trial drug treatment period to avoid viral reactivation; b) For anti-HBc (+), HBsAg (-), anti-HBs ( -) and viral load (-) subjects, do not require prophylactic anti-HBV therapy, but require close monitoring for viral reactivation.

11.Cardiovascular disease meets any of the following: a. Congestive heart failure with cardiac function ≥ NYHA class III; b. Serious arrhythmia requiring drug treatment; c. Acute myocardial infarction, severe or unstable angina pectoris, coronary or peripheral artery bypass, or stenting occurred within 6 months before the first administration; d. Left ventricular ejection fraction (EF) < 60%; e. QTcF interval > 450 ms in men, > 470 ms in women, or risk factors for torsades de pointes such as clinically significant hypokalemia, family history of long QT syndrome, or family history as judged by the investigator History of arrhythmias (eg, pre-excitation syndrome); f. Uncontrolled hypertension (defined as systolic blood pressure ≥150 mmHg and/or diastolic blood pressure ≥100 mmHg after standardized antihypertensive drug treatment).

12.Subjects with active autoimmune disease or a history of autoimmune disease but may relapse, but subjects with the following diseases are not excluded and can be further screened: a. Type 1 diabetes; b. Hypothyroidism (if controllable with hormone replacement therapy alone); c. controlled celiac disease; d. Skin diseases that do not require systemic treatment (eg vitiligo, psoriasis, alopecia); e. Any other disease that will not recur in the absence of external triggers.

13.Subjects with unstable mental illness, alcohol, drug or substance abuse. 14. Female subjects who are pregnant or breastfeeding, or who are expected to become pregnant during the trial period (from the screening visit until 180 days after dosing) and male subjects who are expected to conceive their partner.

15. The adverse reactions of previous anti-tumor therapy have not recovered to (CTCAE 5.0) grade 1 (except for alopecia).

16. The investigator determines that he has a serious uncontrollable disease, or there are other conditions that may affect the acceptance of the treatment in this study, and are considered unsuitable to participate in this researcher.

17. Other investigators deem it unsuitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2021-11-16 (Actual); Primary Completion 2026-06-16 (Estimated); Study Completion 2026-06-16 (Estimated)

PRIMARY OUTCOMES:
MTD (Maximum Tolerance dose) | 2 years
  If ≥2/6 subjects developed DLT, the previous dose group was MTD
DLTs (Dose Limiting Toxicity) | 3 weeks from the first administration
  Toxic reactions according to the NCI-CTCAE 5.0 grading standard that occur within 3 weeks from the first administration, are judged to be drug-related by the investigator, and meet the non-hematological toxicity and hematological toxicity conditions specified in the clinical protocol
Incidence of AE (Adverse Event) and SAE (Serious Adverse Event) | 2 years
  All events with a Grade 3 or above toxicity (defined by the CTCAE v5.0) will be tabulated by event and by relationship to OH2.

SECONDARY OUTCOMES:
OS (Overall Survival) | 2 years
  The overall survival for each patient receiving OH2 will be calculated.
PFS (Progression Free Survival) | 2 years
  Time after OH2 administration to clinical and radiographic disease progression will be evaluated.
Biodistribution and viral shedding | 2 years
  OH2 DNA copy
Immunogenicity | 2 years
  HSV-2 antibody

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zheng Y, Wang X, Ji Q, Fang A, Song L, Xu X, Lin Y, Peng Y, Yu J, Xie L, Chen F, Li X, Zhu S, Zhang B, Zhou L, Yu C, Wang Y, Wang L, Hu H, Zhang Z, Liu B, Wu Z, Li W. OH2 oncolytic virus: A novel approach to glioblastoma intervention through direct targeting of tumor cells and augmentation of anti-tumor immune responses. Cancer Lett. 2024 May 1;589:216834. doi: 10.1016/j.canlet.2024.216834. Epub 2024 Mar 25. PMID 38537773